CLINICAL TRIAL: NCT01081457
Title: Effect of Deep Brain Stimulation on Voluntary and Involuntary Gastrointestinal Motility in Parkinson's Disease
Brief Title: Effect of Deep Brain Stimulation on Gastrointestinal (GI) Motility
Acronym: SCP-Comodig
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Principal Investigator, Guillaume GOURCEROL, MD, University Hospital, Rouen
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 2008/163/HP
Record Dates: First submitted 2010-03-04; First posted 2010-03-05 (Estimated); Last update posted 2012-02-07 (Estimated); Status verified 2012-02

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's disease; deep brain stimulation; GI motility
MeSH Terms: conditions — Parkinson Disease | interventions — Deep Brain Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ON (Active Comparator): Stimulator switched ON
  Interventions: Device: Deep brain stimulation
- OFF (Sham Comparator): Stimulator switched OFF
  Interventions: Device: Deep brain stimulation

INTERVENTIONS:
Device: Deep brain stimulation — Comparison ON vs OFF

SUMMARY:
Parkinson's disease is characterized by extra-pyramidal symptoms as well as digestive involvement with gastrointestinal motility (GI) impairment. Deep brain stimulation has been recently developed as a successful treatment for extrapyramidal symptoms. In addition, preliminary reports suggest that this therapy might be successful to relieve GI symptoms as well. The aim of this study is therefore to assess the effect of deep brain stimulation on GI voluntary as well as involuntary motility.

ELIGIBILITY:
Inclusion Criteria:

* patient over 18 yo
* patient with Parkinson's disease implanted for deep brain stimulation
* patient responders to deep brain stimulation (UPDRS improved by at least 40%)
* patient covered by the french health care system
* patient not taking anti-parkinsonian medication the day before evaluation
* French speaking

Exclusion Criteria:

* patient below 18 yo
* pregnancy
* Severe psychiatric or cognitive disorders
* diabetes mellitus
* morbid obesity
* compulsive eating disorders
* diffuse GI motility impairment (except Parkinson's disease)
* other evolutive neurologic disorders
* previous history of significant GI resection
* inability to swallow or defecate when asked

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2010-01; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Anal pressure | 2 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Rouen University Hospital, Rouen, France

REFERENCES:
- [Derived] Derrey S, Chastan N, Maltete D, Verin E, Dechelotte P, Lefaucheur R, Proust F, Freger P, Leroi AM, Weber J, Gourcerol G. Impact of deep brain stimulation on pharyngo-esophageal motility: a randomized cross-over study. Neurogastroenterol Motil. 2015 Sep;27(9):1214-22. doi: 10.1111/nmo.12607. Epub 2015 Jun 5. PMID 26053217